CLINICAL TRIAL: NCT05144841
Title: A Phase 2 Open-label Clinical Study to Evaluate the Efficacy and Safety of Zilovertamab Vedotin (MK-2140) in Participants With Relapsed or Refractory Diffuse Large B-Cell Lymphoma (waveLINE-004)
Brief Title: A Study to Evaluate Zilovertamab Vedotin (MK-2140) for Relapsed or Refractory Diffuse Large B-Cell Lymphoma (DLBCL) (MK-2140-004)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2140-004; MK-2140-004 (Other: MSD); 2022-501243-33-00 (Registry Identifier: EU CT); U1111-1279-9073 (Registry Identifier: UTN); 2021-003397-32 (EudraCT Number)
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Relapsed or Refractory Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Participants will receive treatment with zilovertamab vedotin 2.5 mg/kg via intravenous (IV) infusion on Day 1 of each 21-day cycle (every 3 weeks (Q3W)) until documented disease progression or any other discontinuation criterion is met.
  Interventions: Biological: MK-2140 (zilovertamab vedotin)
- Arm B (Experimental): Participants will receive treatment with zilovertamab vedotin 2.25 mg/kg via intravenous (IV) infusion on Day 1 of each 21-day cycle (every 3 weeks (Q3W)) until documented disease progression or any other discontinuation criterion is met.
  Interventions: Biological: MK-2140 (zilovertamab vedotin)

INTERVENTIONS:
Biological: MK-2140 (zilovertamab vedotin) — IV infusion of 2.5 mg/kg
  Arms: Arm A
Biological: MK-2140 (zilovertamab vedotin) — IV infusion of 2.25 mg/kg
  Arms: Arm B

SUMMARY:
The purpose of this study is to evaluate zilovertamab vedotin with respect to objective response rate and duration of response per Lugano Response Criteria as assessed by blinded independent central review (BICR). Safety and tolerability will also be evaluated in this Phase 2, single arm, interventional study.

ELIGIBILITY:
Inclusion Criteria:

* Has relapsed or refractory (rr) DLBCL; has progressed after at least 2 lines of prior therapy; and has progressed after auto- stem cell transplant (SCT) or are auto-SCT ineligible. Must have received prior multiagent regimen that includes an alkylating agent. anthracycline, and anti-CD20 (cluster of differentiation 20) monoclonal antibody.
* Has histologically confirmed diagnosis of DLBCL.
* Has radiographically measurable DLBCL per the Lugano Response Criteria.
* Should either be post- chimeric antigen receptor T cell therapy (CAR-T) failure or ineligible for CAR-T (for any reason).
* Life expectancy of at least 3 months.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 assessed within 7 days before time of enrollment.
* Has adequate organ function.

Exclusion Criteria:

* Has received a diagnosis of Primary mediastinal B-cell lymphoma (PMBCL).
* Has undergone solid organ transplant at any time.
* Has a history of any clinically significant cardiovascular conditions within 6 months of screening or serious cardiac arrhythmia requiring medication.
* Has known history of liver cirrhosis.
* Has pericardial effusion or clinically significant pleural effusion.
* Has ongoing Grade >1 peripheral neuropathy.
* Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years.
* Transformed DLBCL from indolent lymphoma.
* In participants with prior allo-SCT, acute graft versus host disease (GVHD) or ongoing evidence of chronic GVHD.
* Has received prior systemic anticancer therapy, including investigational agents within 4 weeks prior to the first dose of study intervention.
* Has received prior radiotherapy within 28 days of start of study intervention. Participants.

must have recovered from all radiation-related toxicities.

* Has ongoing corticosteroid therapy (exceeding 30 mg daily of prednisone equivalent).
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks before the first dose of study intervention.
* Has known active central nervous system (CNS) lymphoma involvement or active CNS involvement by lymphoma.
* Has an active infection requiring systemic therapy.
* Has a known history of human immunodeficiency virus (HIV) infection.
* Has a known history of hepatitis B or known active hepatitis C virus (HCV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-01-08 (Actual); Primary Completion 2026-01-09 (Estimated); Study Completion 2026-01-09 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) per Lugano Response Criteria | Up to approximately 50 months
  ORR is percentage of participants with complete response (CR) or partial response (PR). ORR by cohort, relapsed or refractory (rr) DLBCL as assessed by BICR according to Lugano Response Criteria 2014 in participants treated with zilovertamab vedotin Q3W. CR is the complete radiologic response. PR is a partial response, >=50% decrease in sum of the product of the perpendicular diameters for multiple lesions for up to 6 target measurable nodes and extranodal sites.

SECONDARY OUTCOMES:
Duration of Response (DOR) per Lugano Response Criteria | Up to approximately 50 months
  Duration of Response (DOR) is time from first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first.
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 50 months
  An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience at least one AE will be presented.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 50 months
  An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study treatment due to an AE will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (71):
- United States (19):
  - St. Joseph Hospital-The Center for Cancer Prevention and Treatment ( Site 0229), Orange, California
  - Innovative Clinical Research Institute ( Site 0202), Whittier, California
  - Georgetown University Medical Center ( Site 0204), Washington D.C., District of Columbia
  - Northside Hospital ( Site 0206), Atlanta, Georgia
  - University of Chicago Medical Center ( Site 0207), Chicago, Illinois
  - Franciscan St. Francis Health ( Site 0225), Indianapolis, Indiana
  - University of Maryland-Greenebaum Comprehensive Cancer Center ( Site 0211), Baltimore, Maryland
  - Massachusetts General Hospital-Cancer Center Protocol Office ( Site 0203), Boston, Massachusetts
  - University of Michigan ( Site 0200), Ann Arbor, Michigan
  - Karmanos Cancer Institute ( Site 0216), Detroit, Michigan
  - Saint Louis University Cancer Center ( Site 0209), St Louis, Missouri
  - Atlantic Health System Morristown Medical Center ( Site 0213), Morristown, New Jersey
  - New York Medical College ( Site 0215), Valhalla, New York
  - University of Cincinnati Medical Center-University of Cincinnati Cancer Center ( Site 0217), Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center ( Site 0222), Cleveland, Ohio
  - The James Cancer Hospital and Solove Research Institute at The Ohio State University Comprehensive C, Columbus, Ohio
  - AHN West Penn Hospital ( Site 0212), Pittsburgh, Pennsylvania
  - Avera Cancer Institute- Research ( Site 0233), Sioux Falls, South Dakota
  - MEDICAL COLLEGE OF WISCONSIN ( Site 0234), Milwaukee, Wisconsin
- Princess Margaret Cancer Centre-Division of Medical Oncology and Hematology ( Site 0100), Toronto, Ontario, Canada
- Chile (2):
  - Clínica Alemana de Santiago ( Site 2704), Santiago, Region M. de Santiago
  - James Lind Centro de Investigación del Cáncer ( Site 2705), Temuco, Región de la Araucanía
- China (11):
  - Beijing Cancer hospital ( Site 2900), Beijing, Beijing Municipality
  - SUN YAT-SEN UNIVERSITY CANCER CENTRE-Internal Medicine ( Site 2907), Guangzhou, Guangdong
  - Henan Cancer Hospital-hematology department ( Site 2903), Zhengzhou, Henan
  - Wuhan Union Hospital ( Site 2906), Wuhan, Hubei
  - Hunan Cancer Hospital ( Site 2905), Changsha, Hunan
  - The First Hospital of Jilin University-Hematology ( Site 2910), Changchun, Jilin
  - Fudan University Shanghai Cancer Center ( Site 2908), Shanghai, Shanghai Municipality
  - Shanghai East Hospital ( Site 2902), Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University-Head and Neck Oncology ( Site 2911), Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital-lymphoma ( Site 2901), Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University-Bone marrow transplant centre ( Site 2912), Hangzhou, Zhejiang
- Czechia (2):
  - Fakultní nemocnice Brno Bohunice-Interni hematologicka a onkologicka klinika ( Site 0800), Brno, Brno-mesto
  - Vseobecna fakultni nemocnice v Praze-I. Interní klinika - klinika hematologie ( Site 0801), Prague
- North Estonia Medical Centre Foundation ( Site 0900), Tallinn, Harju, Estonia
- France (2):
  - Centre Hospitalier de la Côte Basque ( Site 1002), Bayonne, Aquitaine
  - Pitie Salpetriere University Hospital-Clinical haematology ( Site 1000), Paris
- Greece (2):
  - Evangelismos General Hospital of Athens ( Site 1214), Athens, Attica
  - General Hospital of Athens "Laiko"-Hematology Department ( Site 1213), Athens, Attica
- Israel (4):
  - Soroka Medical Center-Hematology Department ( Site 1403), Beersheba
  - Shaare Zedek Medical Center ( Site 1404), Jerusalem
  - Hadassah Medical Center ( Site 1402), Jerusalem
  - Sourasky Medical Center ( Site 1400), Tel Aviv
- Italy (4):
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa di Ematologia ( Site 1501), Milan, Lombardy
  - Humanitas-U.O di Oncologia medica ed Ematologia ( Site 1503), Rozzano, Milano
  - IRCCS - AOU di Bologna-Istituto di Ematologia "L. e A. Seragnoli" ( Site 1500), Bologna
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale ( Site 1502), Napoli
- Norway (2):
  - Haukeland Universitetssjukehus ( Site 1601), Bergen, Hordaland
  - Oslo universitetssykehus, Radiumhospitalet ( Site 1600), Oslo
- Poland (5):
  - Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie-Oncology Department ( Site 1707), Krakow, Lesser Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny-Klinika Hematologii, Nowotworow Krwi i Transplantacji Szpiku ( Site, Wroclaw, Lower Silesian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworów Układu Chłonnego ( S, Warsaw, Masovian Voivodeship
  - Szpitale Pomorskie Sp. z o. o.-Hematology and Bone Marrow Transplantation Department ( Site 1702), Gdynia, Pomeranian Voivodeship
  - Pratia Onkologia ( Site 1701), Katowice, Silesian Voivodeship
- South Korea (2):
  - Severance Hospital, Yonsei University Health System-Medical oncology ( Site 0601), Seoul
  - Samsung Medical Center ( Site 0600), Seoul
- Spain (4):
  - Instituto Catalan de Oncologia - Hospital Duran i Reynals-Haematology Department ( Site 2002), L'Hospitalet Del Llobregat, Barcelona
  - Hospital Universitari Vall d'Hebron ( Site 2005), Barcelona
  - Hospital Universitario Fundación Jiménez Díaz-Oncology & Hematology ( Site 2000), Madrid
  - Hospital Universitario de Salamanca - Complejo Asistencial Universitario de Salamanca ( Site 2003), Salamanca
- Sweden (2):
  - Skånes Universitetssjukhus Lund ( Site 2100), Lund, Skåne County
  - Karolinska Universitetssjukhuset Solna ( Site 2102), Solna, Stockholm County
- Thailand (2):
  - Faculty of Medicine Siriraj Hospital ( Site 0701), Bangkok, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital ( Site 0702), Muang, Chiang Mai
- Turkey (Türkiye) (6):
  - Ankara University Hospital Cebeci-hematology ( Site 2300), Ankara
  - Hacettepe Universitesi-Department of Hematology ( Site 2302), Ankara
  - Mega Medipol-Hematology ( Site 2308), Istanbul
  - Dokuz Eylül Üniversitesi-Hematology ( Site 2304), Izmir
  - Ondokuz Mayıs Universitesi ( Site 2306), Samsun
  - Karadeniz Teknik Universitesi Tip Fakultesi-Hematology ( Site 2307), Trabzon

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26167&tenant=MT_MSD_9011